CLINICAL TRIAL: NCT00619437
Title: Genetics of Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Raz Gross, Head, Mental Health Epidemiology, The Gertner Institute for Epidemiology
Other Study IDs: SHEBA-07-4620-RG-CTIL
Record Dates: First submitted 2008-02-10; First posted 2008-02-21 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; genetics; family; multiplex; haplotypes
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cell Lines / DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Genetic etiology in schizophrenia is widely accepted. However, many chromosomal sites were shown to characterize the families of patients with schizophrenia. This is probably due to the high genetic heterogenity of this illness. Thus, it is important to investigate the genetic factor in relatively genetically homogenous populations. Many studies have indicate that Ashkenazy Jews show relative gentic homogenity. Indeed, the genes responsible for most Mendelian disorders of Jewish peoples have been identified. The study will apply genome-wide mutation screening methods to identify candidate allells in subjects of Ashkenazi Jewish ancestry with multiplex schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+;
2. Meet DSM-IV criteria for Schizophrenia;
3. At least one first-degree relative who Meet DSM-IV criteria for Schizophrenia;
4. Can sign the informed consent form.

Exclusion Criteria:

1. Patients suffering from terminal or incurabale disease;
2. Minors, incompetents

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bunzel, MD, Study Director — Psychiatric ward, Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel